CLINICAL TRIAL: NCT02714556
Title: Changes in Ventilation Inhomogeneity and Respiratory Function Following Elective Caesarean Section Under Regional Anaesthesia: a Prospective Observational Study
Brief Title: Changes in Ventilation Inhomogeneity and Respiratory Function Following Elective Caesarean Section Under Regional Anaesthesia
Acronym: VIRCA
Status: Withdrawn | Type: Observational
Why Stopped: Ethical approval not obtained yet as questioning the danger of providing 100% oxygen to parturients.
Sponsor: Walid HABRE (Other)
Responsible Party: Sponsor-Investigator, Walid HABRE, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: VIRCA-2016
Record Dates: First submitted 2016-03-01; First posted 2016-03-21 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy
Keywords: Lung volume; Lung Clearance Index; Functional Residual Capacity; Respiratory function
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Physiologic measures of lung function — Respiratory function tests:
  Nitrogen multiple breath washout (N2MBW) measured with an ultrasonic flowmeter (Exhalyzer D with ICU insert, Eco Medics, Duernten, Switzerland) Forced oscillation technique (FOT) measured with a tremoFlo device (Thorasys, Montreal, Canada)

SUMMARY:
Pregnancy is associated with physiological changes affecting the cardiorespiratory system as a consequence of an increase in both cardiac output and intra-abdominal pressure. The aim of this prospective observational study is to examine the perioperative changes in ventilation inhomogeneity and respiratory function measured by the non-invasive nitrogen multiple breath washout and forced oscillation techniques.

DETAILED DESCRIPTION:
Pregnancy is associated with physiological changes affecting the cardiorespiratory system as a consequence of an increase in both cardiac output and intra-abdominal pressure. These alterations lead to a ventilation/perfusion mismatch which is potentiated by a decrease in functional residual capacity (FRC). These effects explain why pregnant women are more prone to the occurrence of hypoxemia, particularly in the third trimester of their pregnancy. The importance of the ventilation inhomogeneity can be estimated from the lung clearance index (LCI) measured by the non-invasive nitrogen multiple breath washout (N2 MBW) technique. Moreover the loss in lung volume is associated with reduction in respiratory system compliance, which can also be assessed non-invasively by the forced oscillation technique (FOT).

To our knowledge, there is no existing data on LCI or FRC using the aforementioned techniques in pregnant women. Furthermore, existing data on respiratory function in pregnant women is largely restricted to spirometric and body plethysmographic measurements taken primarily in the 1970s-1980s. As such, the important roles of lung ventilation inhomogeneity as well as the potential changes following birth after caesarean section have yet to be completely characterised.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Pregnant woman in the third trimester (37-40 weeks gestational age)
* Scheduled for elective caesarean section under regional (spinal or combined spinal-epidural) anaesthesia

Exclusion Criteria:

* Pregnant women outside 37-40 weeks gestational age
* Non-singleton pregnancy
* Previous history of ≥2 caesarean sections
* History or clinical signs of cardiopulmonary disease in the last 12 months (chronic hypertension, gestational hypertension, preeclampsia, asthma, acute or chronic bronchitis, others)
* Positive current smoking status
* Pre-pregnant body mass index (BMI) >30 kg/m2 (based on booking records)
* Respiratory infection <2 weeks prior to surgery
* Inability to perform the respiratory function tests

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women scheduled for elective caesarean section in gestational weeks 37-40
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Perioperative changes in ventilation inhomogeneity (LCI) following delivery by caesarean section | 1-3 days prior to caesarean section until 5 days postoperative
  Nitrogen multiple breath washout technique

SECONDARY OUTCOMES:
Alterations in FRC throughout the postpartum period | 1-3 days prior to caesarean section until 5 days postoperative
  Nitrogen multiple breath washout technique
Changes in respiratory mechanics: respiratory system compliance (Crs) | 1-3 days prior to caesarean section until 5 days postoperatively
  Forced oscillation technique
Changes in respiratory mechanics: airway resistance (Raw) | 1-3 days prior to caesarean section until 5 days postoperatively
  Forced oscillation technique
Perioperative respiratory complications | During caesarean section until 5 days postoperatively
  Apnoea/bradypnoea, oxygen desaturation <90%/hypoxemia, hypoventilation/atelectasis, pulmonary embolism, incoercible cough
Perioperative respiratory interventions | During caesarean section until 5 days postoperatively
  Intubation, oxygen therapy, bronchodilator, adrenaline, continuous positive airways pressure (CPAP), respiratory physiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Walid Habre, MD, PhD, Study Director — University of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No